CLINICAL TRIAL: NCT04367545
Title: Development of a Molecular Diagnostic Strategy for SARS-CoV2 Based on Saliva in the Context of the COVID-19 Pandemic
Acronym: MolCOVID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020/0094/OB
Record Dates: First submitted 2020-04-27; First posted 2020-04-29 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: COVID; RT-ddPCR Multiplex

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient with COVID-19 infection suspicion (Experimental): Patient with COVID-19 infection suspicion are tested using standard diagnosis method
  Interventions: Diagnostic Test: Saliva collection

INTERVENTIONS:
Diagnostic Test: Saliva collection — Saliva collection will be done in addition to standard diagnosis collection (nasopharyngeal collection using swab)

SUMMARY:
The objective of the study is to develop and validate a molecular diagnostic strategy (RT-ddPCR multiplex) of COVID-19 based on a saliva sample and alternative to the RT-qPCR method, in order to :

1. to compensate for the risk of a shortage of diagnostic kits, reagents and materials necessary for molecular diagnosis;
2. to increase the molecular diagnostic capacity of COVID-19 at the Rouen University Hospital;
3. and to have a method compatible with screening extended to populations at risk.

ELIGIBILITY:
Inclusion Criteria:

* Person aged over 18 years presenting to the COVID-19 consultation of the Rouen University Hospital for screening
* Person affiliated to a social security scheme

Exclusion Criteria:

* Person objecting to participation in the research after reading information
* Person under the protection of justice,
* Person deprived of their liberty by administrative or judicial decision (guardianship, curatorship, etc.)
* Patient under guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2020-04-16 (Actual); Primary Completion 2020-05-17 (Actual); Study Completion 2020-05-17 (Actual)

PRIMARY OUTCOMES:
Number of positive patient using saliva method compared to number of positive patient using standard method | One hour
Number of negative patient using saliva method compared to number of negative patient using standard method | One hour

CONTACTS AND LOCATIONS:
Overall Officials: Thierry FREBOURG, Pr, Principal Investigator — University Hospital, Rouen
Locations (1):
- Rouen University Hospital, Rouen, France

IPD SHARING:
Plan to Share IPD: No